CLINICAL TRIAL: NCT03699410
Title: A Proof-of-concept, Prospective, Observational Study to Investigate the Value of Liquid Biopsies to Predict Tumor Response After Neoadjuvant Chemo-radiotherapy in Patients With Locally Advanced Rectal Cancer: the LiBReCa Study
Brief Title: Observational Study on Rectal Cancer to Verify if Response After Chemo-radiotherapy Can be Predicted With a Particular Blood Test.
Acronym: LiBReCa
Status: Terminated | Type: Observational
Why Stopped: failure to identify complete responders since ctDNA disappears after radiotherapy in most patients.
Sponsor: Dimitri Christoforidis (Other)
Collaborators: Clinical Trial Unit Ente Ospedaliero Cantonale (Other)
Responsible Party: Sponsor-Investigator, Dimitri Christoforidis, Deputy Chief of the Surgery and Visceral Surgery Departments, Ente Ospedaliero Cantonale, Bellinzona
Organization: Ente Ospedaliero Cantonale, Bellinzona (Other)
Other Study IDs: ORL-CHIR-002
Record Dates: First submitted 2018-10-05; First posted 2018-10-09 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-10

CONDITIONS: Locally Advanced Rectal Cancer
MeSH Terms: interventions — Neoadjuvant Therapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue: the biopsy at the time of diagnosis will be characterized using next-generation sequencing (NGS).
  Blood: circulating tumor DNAs (ctDNAs) from plasma collected at diagnosis and at various time-points in the patients' treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Neoadjuvant radiotherapy — Radiotherapy with total dose of at least 50 Gy on the tumor (cT) and the involved nodes (cN+) and with standard fractionation (1.8 Gy/fraction), 5 days/week.
Drug: Neoadjuvant chemotherapy — Oral Capecitabine, at the standard dose of 825 mg/m2 twice daily, concomitant to radiotherapy.
Procedure: Radical surgery — The time point of surgery is usually dependent on surgeon's and institutional habits and lies within 6 to 12 weeks after the end of nCRT. Surgeons participating in this study will be asked to operate patients on the 10th week after the end of nCRT.

SUMMARY:
Research project for patients with locally advanced rectal cancer in which biological material and health-related personal data are collected.

The aim is to investigate if an additional method (liquid biopsies) can predict the response after chemo-radiotherapy and before surgery.

DETAILED DESCRIPTION:
The standard treatment for locally advanced rectal cancer (T3 -T4 and / or N+) is neoadjuvant (pre-operative) chemo-radiotherapy (nCRT) followed by radical surgery. In patients after complete response following nCRT, surgery may not add any survival benefit but it is still performed.

Since clinical complete response has only partial concordance with pathological complete response, an additional method that helps identify those patients with a true complete response is needed to avoid unnecessary surgery and its associated potential complications..

The hypothesis underlying this study is that the quantitative and qualitative evaluation of circulating tumor DNA (ctDNA) of liquid biopsy, based on the amount of ctDNA or on the detection of specific gene alterations respectively, may be directly correlated to the clinical, histopathological and radiological response of the tumor to nCRT.

This study will not interfere with the patient's routine treatment pathway and there will be no deviation from the standard of care. The only additional study intervention will be the collection of blood samples at 6 different time points which can be combined with the regular blood examination performed during the treatment.

At the time of diagnosis, tumor staging and histopathology on tumor biopsy will be performed. Patients will receive standardized neoadjuvant therapy and will be operated after an observational period of 10 weeks. Peripheral blood sample will be collected at 6 time points: pre-nCRT, at the end of the nCRT, at 4th and 7th week post-CRT, on the day of the surgery (before surgical resection), on the post-operative day 5 (in hospital). Mesenteric blood sample will be collected intra-operatively on the day of the surgery. Tumor sampling will be performed during tumor staging, as standard of care, and on the resection specimen. A combined qualitative and quantitative approach for the molecular characterization of tissue and liquid biopsy using next-generation sequencing will be carried out.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Locally advanced rectal cancer (T3 or T4, and/or N+) requiring long course nCRT (as decided by the regional tumor board)
* Patient fit for surgery and treated with curative intent
* Willingness to complete all clinical and radiological examinations foreseen by the study
* Availability of tissue specimen for molecular characterization at baseline
* Written informed consent

Exclusion Criteria:

* Presence of metastases
* Insufficient material on the tissue biopsy to be left in archives of the Cantonal Institute of Pathology for further evaluations/analyses
* Insufficient amount of tumor cells in the tissue biopsy for the molecular characterization
* Inability to consent and follow the procedures of the study
* Women who are pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with locally advanced rectal cancer afferent to participating sites
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2018-08-28 (Actual); Primary Completion 2020-10-20 (Actual); Study Completion 2020-10-20 (Actual)

PRIMARY OUTCOMES:
Negative Prognostic Value (NPV) | day of surgery
  NPV of the liquid biopsy of ctDNA drawn from the mesenteric and peripheral blood

CONTACTS AND LOCATIONS:
Overall Officials: Dimitri Christoforidis, Principal Investigator — Surgery and Visceral Surgery Departments Regional Hospital of Lugano
Locations (2):
- Switzerland (2):
  - Regional Hospital of Lugano, Lugano
  - Clinica Luganese Moncucco, Lugano